CLINICAL TRIAL: NCT05880849
Title: Testing Whether Choline Normalizes Lipid Metabolism in APOE4 Carriers
Brief Title: Choline Effects - Pre-symptomatic AD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Paul E Schulz (Other)
Collaborators: M.D. Anderson Cancer Center (Other); Massachusetts Institute of Technology (Other); Balchem Corporation (Industry)
Responsible Party: Sponsor-Investigator, Paul E Schulz, Professor, Department of Neurology, The University of Texas Health Science Center, Houston
Organization: The University of Texas Health Science Center, Houston (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-22-0637
Record Dates: First submitted 2023-05-10; First posted 2023-05-30 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Alzheimer Disease
Keywords: pre-symptomatic AD
MeSH Terms: conditions — Alzheimer Disease | interventions — Choline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Choline (Experimental): 2.2 g of choline, given as choline bitartrate, for a total of 180 days.
  Interventions: Drug: Choline

INTERVENTIONS:
Drug: Choline — Eight 275mg capsules taken orally twice daily (4 capsules with breakfast & 4 capsules with dinner) x 180 days
  Other Names: Choline Bitartrate; VitaCholine(R)

SUMMARY:
The purpose of this study is to test the safety, tolerability, and effects of choline in people with increased risk of Alzheimer's Disease (AD), also known as pre-symptomatic AD. Choline is a dietary supplement, but is being investigated to see if it has any effects on the progression to AD.

DETAILED DESCRIPTION:
The purpose of this study is to determine the safety and tolerability, as well as the biochemical effects of choline bitartrate over a 6-month treatment period in a moderately sized population harboring at least one copy of the APOE4 gene. APOE is a protein involved in lipid transport. Studies show that the APOE4 variant is strongly associated with an increased risk of Alzheimer's Disease. It is unclear how APOE4 results in an increased risk for AD, but a recent study identified a novel molecular pathway, which showed that APOE4-induced dysfunction of lipid metabolism in neurons by cellular accumulation of unsaturated lipids. The investigators hypothesize that choline supplementation normalizes the APOE4-mediated dysregulation by normalizing the Kennedy pathway in neuronal cells, thus stabilizing the lipid metabolism and concomitantly restoring normal cell function by increasing phosphatidylcholine activity via the Kennedy pathway. To evaluate this, the investigators will test if choline supplementation will decrease the ratio of unsaturated lipids to saturated lipids (the fatty acid desaturation index) in cerebrospinal fluid by 15% and increase phosphatidylcholine by 100%.

ELIGIBILITY:
Inclusion Criteria:

1. Has signed an informed consent form before any assessment is performed as part of the study.
2. Be male or female between 55 and 80 years old.
3. Be able to understand the nature of the study and have the opportunity to have all questions answered.
4. Has tested positive for at least one copy of ApoE4.
5. Has an MMSE score of 24 or greater. (can be based on documented result obtained within the previous 3 months).
6. Is in the opinion of the Investigator, in good general medical health based upon medical history, physical examination, laboratory tests, vital signs and EKG.
7. Has normal levels of Homocysteine in blood tests. A normal blood level is between 5 to 15 micromoles (mcmol/L)
8. Completes the dietary interview with dietician.
9. Females must be considered post-menopausal or not of child bearing potential.

Exclusion Criteria:

1. Current medical or neurological condition that might impact cognition or performance on cognitive assessments. (e.g. TBI, Parkinson's disease, multiple sclerosis, etc.)
2. Inability or unwillingness of patient to undergo neuropsychological testing.
3. Advanced, severe progressive or unstable disease that may interfere with the safety, tolerability and study assessments, or put the participant at special risk. (e.g. significant cardiac disease, severe renal impairment, severe hepatic impairment etc.)
4. History of malignancy of any organ system, treated or untreated, within the past 60 months.
5. Inability or unwillingness to undergo Lumbar Punctures.
6. High dietary choline intake (more than 450mg) as determined by dietician
7. Any condition, which in the opinion of the investigator, would put the subject at undue risk or would interfere with evaluation of the investigational product or interpretation of subject safety or study results.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-06-26 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-10-10 (Actual)

PRIMARY OUTCOMES:
Changes in the fatty acid desaturation index (FADI) in the CSF following choline supplementation | baseline, 6 months
  FADI will be utilized to determine whether unsaturated to saturated lipids decreases by 15%
Changes in phosphatidylcholine (PC) in the CSF following choline supplementation | baseline, 6 months
  FADI ( fatty acid desaturation index) will be utilized to determine whether saturated PC increases by 100%

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events | 9 months
  Safety endpoints will be monitored throughout the study and number of incidents reported at end of study. Aggregate values and percentages will be reported
Changes in phospholipids in CSF following choline supplementation | Baseline and 6 months
  Will compare scaled intensity between baseline and 6 months.
Changes in phosphatidylcholine in blood following choline supplementation | Baseline and 6 months
  Aggregate values and percentages will be reported.
Changes in choline in blood following choline supplementation | Baseline and 6 months
  Aggregate values and percentages will be reported
Changes in proinflammatory cytokines in blood plasma following choline supplementation | Baseline and 6 months
  Proinflammatory cytokine panel in plasma will be measured using commercially available immunosorbent assays to determine potential treatment effects. Aggregate values and percentages will be reported. Each sample will be tested in triplicate.
Changes in neurofilament light chain (Nf-L) in CSF following choline supplementation | Baseline and 6 months
  Levels of NfL in CSF will be measured using commercially available immunosorbent assays to determine potential treatment effects. Aggregate values and percentages will be reported. Each sample will be tested in triplicate.
Changes in amyloid-β 42/40 ratio CSF following choline supplementation | Baseline and 6 months
  Levels of amyloid-β 42/40 ratio in CSF will be measured by LC/MS/MS assays. Aggregate values and percentages will be reported.
Changes in p-Tau/Total Tau ratio in CSF following choline supplementation | Baseline and 6 months
  Levels of p-Tau/Total Tau will be measured by LC/MS/MS assays. Aggregate values and percentages will be reported.

OTHER OUTCOMES:
Change in Mini-Mental Status Examination (MMSE) following choline supplementation | Baseline and 6 months
  Cognition measured by MMSE. Scoring: 24-30 no cognitive impairment; 18-23 mild cognitive impairment; 0-17 severe cognitive impairment.
Change in Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) scores following choline supplementation | Baseline and 6 months
  Cognitive decline measured by RBANS. Total Score subtest ranges: List Learning (0-40); Story Memory (0-24); Figure Copy (0-20); Line Orientation (0-20); Picture Naming (0-10); Semantic Fluency (4-40); Digit Span (0-16); Coding (0-89); List Recall (0-10); List Recognition (0-20); Story Recall (0-12); Figure Recall (0-20). Use Stimulus Booklet to convert Total Scores to Index Scores and Sum of Index Scores to Total Scale. Total Scores can range from 40 to 160. The RBANS scores are displayed as standard scores with means of 100 and a standard deviation of 15. Average/Mild Impairment (standard scores of 70 or above), Moderate Impairment (standard scores from 55 to 69), and Severe Impairment (standard scores <54).
Change in Functional Activities Questionnaire (FAQ) scores following choline supplementation | Baseline and 6 months
  Measure instrumental activities of daily living (IADLs) by FAQ. Sum scores (range 1-30). Cut-point of 9 (dependent in 3 or more activities) is recommended to indicate impaired function and possible cognitive impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Paul E Schulz, MD, Principal Investigator — The University of Texas Health Science Center at Houston (UTHealth)
Locations (1):
- The University of Texas Health Science Center at Houston (UTHealth), Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No